CLINICAL TRIAL: NCT06186518
Title: Impact of the PIKSEC App on Intravenous Insertion Success, Pain, and Emotional Manifestation in Pediatric Patients: a Non-Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Yeliz Taşdelen, Registered Nurse, RN, Zonguldak Bulent Ecevit University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: BEU-YTASDELEN-002
Record Dates: First submitted 2023-12-05; First posted 2024-01-02 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-05

CONDITIONS: Nurse's Role; Peripheral Venous Catheterization; Pain; Emotional Stress
MeSH Terms: conditions — Pain; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The study will be conducted in the pediatric clinic of a training and research hospital. Initially, control group data will be gathered through the routine peripheral intravenous catheter placement practices within the service. Subsequently, data for the experimental group will be collected using the PİKSEÇ application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other)
  Interventions: Other: Routine care
- PİKSEÇ group (Experimental)
  Interventions: Other: PİKSEÇ

INTERVENTIONS:
Other: PİKSEÇ — In designing the PİKSEÇ application, the Turkish validity and reliability version of the 'Difficult Intravenous Access Score' and a literal translation of the miniMAGIC instructions were utilized. The application serves as a guideline for nurses during peripheral intravenous catheter insertion, taking into account parameters such as the patient's age, urgency status, anxiety, and vein characteristics, providing tailored suggestions.
  By utilizing the application, nurses can follow evidence-based guidelines more efficiently, ensuring a faster and more practical adherence to the PIVC intervention procedure, ultimately contributing to a safer peripheral intravenous catheter insertion process.
  Arms: PİKSEÇ group
Other: Routine care — The pediatric unit's PIVC insertion process will be routinely performed in routine care.
  Arms: Control group

SUMMARY:
The study employed a post-test non-randomized controlled trial to assess the impact of the PİKSEÇ (Peripheral Intravenous Catheter Selection) application on the success of peripheral intravenous catheter (PIVC) placement, as well as on the pain and emotional level scores of hospitalized preschool children aged 3-6 years. In preschool children, aged 3-6 years, who were hospitalized, anxiety about losing body integrity is commonly observed. Children tend to think that all the material inside their bodies can come out through a wound or hole during invasive procedures. Therefore, it becomes crucial to reduce anxiety related to invasive procedures in children of this age group. In this context, the study aimed to be conducted in preschool children.

ELIGIBILITY:
Inclusion Criteria:

* Being a child in the 3-6 age group
* PIVC to be inserted
* Parents volunteering their child to participate in the study and signing the consent form
* Parents are literate

Exclusion Criteria:

* Physical and mental disabilities,
* The parent has an obstacle to communication (being mentally stable, etc.)

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
PIVC success rate at first insertion | From the day the first sample was included in the study to the day the last sample was included, an estimated 4 months.
Number of PIVC attempts | Starts with the first PIVC attempt in each sample and ends with the successful PIVC attempt, an estimated 15 minutes.. Can be between 1 and 4 attempts.
PIVC attempts duration | Measured with a stopwatch for 4 months.
  It starts with the attachment of the tourniquet during the first PIVC attempt and ends with the fixation of the PIVC.
Wong-Baker Faces Pain Rating Scale Score during PIVC attempt | It starts with the attachment of the tourniquet during the first PIVC attempt and ends with the fixation of the PIVC, an estimated 2 minutes.
  The Wong-Baker Faces Pain Rating Scale has a minimum score of 0 and a maximum score of 5. An increase in score means an increase in pain.
Emotional Indicators Scale in Children Score during PIVC attempt | It starts with the attachment of the tourniquet during the first PIVC attempt and ends with the fixation of the PIVC, an estimated 2 minutes..
  The scale has a minimum score of 5 and a maximum score of 25. An increase in the score indicates a worsening of the emotional state.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük Educational and Research Hospital, Karabük, Center, Turkey (Türkiye)